CLINICAL TRIAL: NCT05860452
Title: Effectiveness of TAP (Transversus Abdominis Plane) Block for Postoperative Pain Relief After Abdominal Aortic Surgery
Brief Title: Effectiveness of TAP (Transversus Abdominis Plane) Block for Abdominal Aortic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Gordan Mijovski, assist.dr.Gordan Mijovski dr. med., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAP study
Record Dates: First submitted 2023-04-23; First posted 2023-05-16 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Abdominal Aortic Aneurysm; Abdominal Aortic Stenosis; Syndrome, Leriche
Keywords: Abdominal aorta, TAP
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Leriche Syndrome | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Dedicated anaesthetic nurse will prepare the syringes for administering the TAP block for each participant. She will be the only person to know which group each participant has been allocated to. Since local anaesthetic and normal saline have no color the anaesthetist performing the block will be, as will the doctors and nurses in postoperative care, blinded to the group each participant has been allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ropivacaine (Active Comparator): Participants in this group will receive TAP block with 0,75%, bilaterally.
  Interventions: Other: ropivacaine
- normal saline (Placebo Comparator): Participants in this group will receive TAP block with normal saline, bilaterally.
  Interventions: Other: normal saline

INTERVENTIONS:
Other: ropivacaine — single shot bilateral TAP block
  Arms: ropivacaine
Other: normal saline — single shot bilateral TAP block
  Arms: normal saline

SUMMARY:
The goal of this study is to learn about the effectiveness of TAP block for pain relief after vascular surgery on the abdominal aorta.

The main question the investigators are looking to answer is whether the TAP block lowers the dose of opioid required after abdominal aortic surgery.

DETAILED DESCRIPTION:
The surgery on the abdominal aorta requires extended haemodynamic monitoring and is performed under general anaesthesia. After applying general anaesthesia, the patients will receive a TAP block (subcostal approach) before the start of the surgery.

During the procedure the patients will receive both opioid and nonopioid analgesics, as part of the standard perioperative protocol for abdominal aortic surgery.

After the procedure all patients will receive following the standard protocol for pain relief after abdominal aortic surgery - NSAIDs and nonopioid analgesics regularly. All patients will postoperatively receive opioid as a rescue drug as needed (PCA).

Participants will be randomly allocated in two groups, where one group will receive local anaesthetic for the TAP block and the control group will receive normal saline for the TAP block. The anaesthetist, the nurses and doctors in the postoperative care will all be blinded as to the group in which each patient is allocated.

The participants will be followed from surgery until discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted for an elective vascular surgery on abdominal aorta that agree and give written consent to be included in the study.

Exclusion Criteria:

* Patients allergic to the drugs we will use in the study, local anaesthetic, nonopioid analgesics, NSAIDs.
* Patients with pain syndromes that are preoperatively already on any kind of chronic pain therapy.
* Patients that will experience surgical complications that requires reoperation will be excluded postoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Cumulative dose of opioid in the first 48 hours after surgery | 48 hours after surgery
  Cumulative dose of opioid, administered in the first 48 hours after surgery

SECONDARY OUTCOMES:
Length of hospital stay | up to 2 weeks
  Length of hospital stay after surgery measured in days
Patient satisfaction with pain relief | up to 7 days postoperatively
  The participants will be asked to grade their satisfaction of pain relief on a 5 rating satisfaction scale from 1 - 5 (where 1 is best and 5 is worst).
  1.very satisfied 2.satisfied 3. neither satisfied nor dissatisfied 4.dissatisfied 5. very dissatisfied
Return of peristalsis | up to 2 weeks
  Return of peristalsis after surgery measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Gordan Mijovski, MD, Principal Investigator — UMC Ljubljana
Locations (1):
- UMCLjubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No